CLINICAL TRIAL: NCT04840615
Title: Phase I Study of Intratumor Injection of Anti-Mesothelin Immunotoxin LMB-100 With Ipilimumab in Malignant Mesothelioma
Brief Title: Intratumor Injection of Anti-Mesothelin Immunotoxin LMB-100 With Ipilimumab in Malignant Mesothelioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was closed early due to slow accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raffit Hassan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000059; 000059-C
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Mesothelioma
Keywords: Immunotherapy; Checkpoint Inhibitor; anti CTLA-4
MeSH Terms: conditions — Mesothelioma | interventions — LMB-100; Ipilimumab; Diphenhydramine; Famotidine; Acetaminophen; Dexamethasone; Calcium Dobesilate; Biopsy; Magnetic Resonance Imaging; Electrocardiography; Echocardiography; Caves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Intra-tumoral LMB-100 Administration (Experimental): Those with pleural or peritoneal mesothelioma receiving intra-tumoral administration of LMB-100 + ipilimumab for up to 4 cycles.
  Interventions: Biological: LMB-100; Drug: ipilimumab; Drug: Diphenhydramine; Drug: Famotidine; Drug: Acetaminophen; Drug: Dexamethasone; Procedure: Biopsy; Diagnostic Test: FDG-PET; Diagnostic Test: CT CAP; Diagnostic Test: MRI; Diagnostic Test: ECG; Diagnostic Test: Echocardiogram

INTERVENTIONS:
Biological: LMB-100 — LMB-100 administered into lesion on days 1 and 4 during cycle 1.
Drug: ipilimumab — Administered intravenously once per cycle up to three 21-day cycles. Administration will occur during cycles 2,3,4.
  Other Names: Yervoy
Drug: Diphenhydramine — Infusion related reactions precaution: All participants will be premedicated with 25-50 mg Diphenhydramine by mouth (PO) or intravenous (IV) (or alternative antihistamine at adequate dose) 30-60 minutes (+ 30 minutes) prior to each LMB-100 administration.
  Other Names: Benadryl
Drug: Famotidine — Infusion related reactions precaution: All participants will be premedicated with 20 mg Famotidine by mouth (PO) or intravenous (IV) (or alternative histamine H2- receptor antagonists (H2) blocker at adequate dose) 30-60 minutes (+ 30 minutes) prior to each LMB-100 administration.
  Other Names: Pepcid
Drug: Acetaminophen — Infusion related reactions precaution: All participants will be premedicated with 650 mg Acetaminophen by mouth (PO) or intravenous (IV) 30-60 minutes (+ 30 minutes) prior to each LMB-100 administration.
  Other Names: Tylenol
Drug: Dexamethasone — Additional infusion precaution at infusions of LMB-100 after Cycle 1 Day 1 (as appropriate): Dexamethasone 20 mg by mouth (PO), 6-12 hours prior to LMB-100 administration OR 10mg, intravenous (IV), 30-60 minutes prior to LMB-100 administration OR equivalent dose of another corticosteroid as clinically indicated.
  Other Names: Ozurdex
Procedure: Biopsy — As feasible at screening, Cycle 1 Day 1 and 5, Cycle 2, 3, & 4 Day 1, and Cycle 4 Day 21 (±7 days).
Diagnostic Test: FDG-PET — At screening, at the end of cycles 2 & 4 ± 7 days, Follow-Up Visit (4-6 weeks after end of treatment), and Long-Term Follow-Up (every 6-12 weeks).
  Other Names: Fluorodeoxyglucose-positron emission tomography
Diagnostic Test: CT CAP — At screening, at the end of cycles 2 & 4 ± 7 days, Follow-Up Visit (4-6 weeks after end of treatment), and Long-Term Follow-Up (every 6-12 weeks).
  Other Names: Computed tomography of the chest, abdomen and pelvis
Diagnostic Test: MRI — At screening, at the end of cycles 2 & 4 ± 7 days, Follow-Up Visit (4-6 weeks after end of treatment), and Long-Term Follow-Up (every 6-12 weeks).
  Other Names: Magnetic resonance imaging
Diagnostic Test: ECG — At screening, Cycle 1 Day 1, Cycles 2, 3, & 4 Day 1 and Follow-Up Visit (4-6 weeks after end of treatment).
  Other Names: Electrocardiogram
Diagnostic Test: Echocardiogram — At screening.
  Other Names: Echo

SUMMARY:
Background:

Mesothelioma is a type of cancer. It originates in cells that line human body cavities. Most people have advanced disease when they are diagnosed. Researchers want to see if a combination of drugs can help.

Objective:

To find a safe dose of LMB-100 in combination with ipilimumab when LMB-100 is injected into tumors.

Eligibility:

Adults ages 18 and older with malignant pleural or peritoneal mesothelioma, that cannot be cured with surgery and has not responded to standard first-line treatments for mesothelioma.

Design:

Participants will be screened with:

* Tumor biopsy or effusion, if needed
* Medical history
* Physical exam
* Blood and urine tests
* Imaging scans
* Heart and lung function tests
* Pregnancy test, if needed

Some screening tests will be repeated during the study.

Participants will get LMB-100 on Days 1 and 4 for up to 2 cycles. Each cycle lasts 21 days. They will stay in the hospital for about 8 days each time they get LMB-100. It will be injected into their tumor with needles.

Participants will get ipilimumab through a tube that is put in a vein. It will be given on Day 2 of the first 2 cycles and Day 1 of the next 2 cycles.

Participants will be assessed for how well they do daily activities. They will give blood and tissue samples for research.

Participants will have a safety visit 4 to 6 weeks after the last dose of the study drugs. Then they will have scans every 6 weeks until their disease gets worse. If their tumor gets bigger, they will have phone, video, or email follow-ups every 12 weeks.

Participants will be on this study for life....

DETAILED DESCRIPTION:
Background:

LMB-100, and a closely related immunotoxin, SS1P, also targeting mesothelin, given intravenously, have been studied in Phase 1 clinical studies for mesothelioma and pancreatic cancer.

LMB-100 given intravenously results in systemic inflammation in patients, but as a single agent has limited anti-tumor efficacy.

Almost all patients develop neutralizing anti-LMB-100 antibodies after 2 cycles of therapy.

Intra-tumoral delivery of LMB-100 has been shown to induce immune cell infiltration in immune-competent mice, bearing murine malignant mesothelioma tumors. Combination with cytotoxic T-lymphocyte associated protein 4 (CTLA-4) blockage eradicates murine tumors by promoting anti-cancer immunity.

Ipilimumab is a fully human anti CTLA-4 monoclonal antibody, that is approved for treatment of melanoma and in combination with nivolumab for many solid tumors.

It is hypothesized that intra-tumoral delivery of anti-mesothelin immunotoxin LMB-100 in combination with ipilimumab will result in greater anti-tumor efficacy in patients with mesothelioma.

Objective:

To determine the safety and feasibility of intra-tumoral LMB-100 injection plus ipilimumab infusion in patients with mesothelioma

To identify the recommended phase 2 dose (RP2D) of intratumorally administered LMB-100 + ipilimumab in patients with malignant mesothelioma

Eligibility:

Histologically confirmed pleural or peritoneal mesothelioma not amenable to potentially curative surgical resection.

Have locally accessible disease suitable for intra-tumor injection of LMB-100. This includes superficial or visceral lesions.

Subjects must have received prior immune checkpoint therapy with anti-Programmed cell death protein 1 (PD-1)/Programmed death-ligand 1 (PD-L1) inhibitors alone or in combination with anti-CTLA4 blocking antibodies, as well as platinum-based chemotherapy.

Age >= 18 years.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Adequate organ and bone marrow function

Subjects with clinically significant pericardial effusion are excluded.

Chemotherapy within 3 weeks or radiotherapy within 2 weeks prior to start of study therapy, is prohibited.

Subjects with active central nervous system (CNS) metastasis are excluded.

Subjects with active autoimmune disease for which they have received systemic immunosuppressive medications during the previous 2 years (excluding daily glucocorticoid-replacement therapy for conditions such as adrenal or pituitary insufficiency) are excluded.

Subjects with active interstitial lung disease, or a history of pneumonitis or interstitial lung disease for which they had received glucocorticoids are excluded.

Design:

This is an open-label, single center phase I dose escalation study of intratumorally administered LMB-100 followed by ipilimumab in subjects with malignant mesothelioma.

Subjects will receive intratumorally administered LMB-100, beginning at dose level 1, in 21-day cycles. LMB-100 will be given on days 1 and 4 of cycle 1, and ipilimumab is given on day 1 of cycles 2-4.

Tumor biopsies will be performed prior to each administration of LMB-100, on day 1 of cycle 2 and after completion of ipilimumab therapy to evaluate changes in the tumor immune microenvironment.

Up to 14 evaluable subjects will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histologically confirmed malignant pleural or peritoneal mesothelioma not amenable to potentially curative surgical resection. The diagnosis will be confirmed by the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI).
  2. Tumor must have epithelioid histology determined by the Laboratory of Pathology at the NCI. If the patient has biphasic histology, the epithelioid component must be >50%
  3. Have provided archival tumor tissue sample or able to provide newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred, to slides. Newly obtained biopsies are preferred to archived tissue.

     Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
  4. Have disease locally, accessible disease to suitable for intra-tumoral injection of LMB- 100.
  5. Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
  6. Subjects must have received prior immune checkpoint therapy with anti-Programmed cell death protein 1 (PD-1)/Programmed death-ligand 1 (PD-L1) inhibitors alone or in combination with anti-CTLA4 blocking antibodies, as well as platinum-based chemotherapy.
  7. Age >= 18 years.
  8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Evaluation of ECOG is to be performed within 28 days prior to initiation of study therapy.
  9. Have adequate organ and marrow function as defined below:

     System and Laboratory Value

     Hematological -

     hemoglobin >= 9 g/dL(a)

     absolute neutrophil count >= 1,500/mcL

     platelets >= 100,000/mcL

     Hepatic

     total bilirubin <= 2.5 X institutional upper limit of normal (ULN) OR direct bilirubin <=ULN for participants with total bilirubin levels >1.5 X ULN

     Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 X institutional ULN (<= 5 X ULN for participants with liver metastases)

     Renal

     Creatinine <=1.5 x ULN OR Measured or calculated(b) creatinine clearance (glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl) >= 50 mL/min for participant with creatinine levels; > 1.5 X institutional ULN

     Coagulation

     International normalized ratio (INR) OR prothrombin time (PT); Activated partial thromboplastin time (aPTT): <=1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT, is within therapeutic range of intended use of anticoagulants

     ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.
     1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
     2. Creatinine clearance (CrCl) should be calculated per institutional standard.
  10. Must have left ventricular ejection fraction >50%.
  11. The effects of LMB-100 on the developing human fetus are unknown. For this reason and because ipilimumab is a Category C agent, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) while on study therapy and for four months after the last dose of study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  12. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 3 weeks prior to initiation of study therapy.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 3 weeks after the last dose of the previous investigational agent. Patients with active devices will be excluded from the study.
2. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to initiation of study therapy.
3. Has active systemic issues as bleeding diathesis or active infections
4. Presence of a clinically significant pericardial effusion
5. Has severe hypersensitivity (>=Grade 3) anti-CTLA4 therapies and/or any of their excipients.
6. Has received prior radiotherapy to the site of local administration
7. Subjects who have received LMB-100 previously
8. Has received prior systemic anti-cancer therapy including investigational agents within 3 weeks prior to initiation of study therapy. Patients who have received prior anti-PD-1/PD- L1 or CTLA4 antibodies are eligible. Any toxicity related to these agents must have resolved to grade 1 and they must not be on systemic immunosuppressive therapies (physiologic dose of steroids are permitted).
9. Has received prior radiotherapy to site other than target lesion within 2 weeks prior to initiation of study therapy. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (<=2 weeks of radiotherapy) to non-CNS disease.
10. Has not recovered from all adverse events (AEs) due to previous therapies to <=Grade 1 or baseline. Participants with <=Grade 2 neuropathy may be eligible. If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to initiation of study therapy.
11. Has received a live vaccine within 30 days prior to initiation of study therapy. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist(R)) are live attenuated vaccines and are not allowed.
12. Is receiving therapeutic anti-coagulation. Patients receiving prophylactic anticoagulation may be eligible if in the opinion of the study team, anti-coagulation may be stopped during the time of LMB-100 administration and tumor biopsies.
13. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to initiation of study therapy.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has a QT corrected for heart rate by Fridericia's cube root formula (QTcF) interval >480 milliseconds.
16. Has a history of (non-infectious) pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject s participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. A woman of childbearing potential who has a positive pregnancy test within 72 hours prior to initiation of study therapy. If the using a urine test and test positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event, that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative, in order for subject to start receiving study medication.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 4 months after the last dose of trial treatment. Pregnant women are excluded from this study because LMB-100 + ipilimumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMB-100 + ipilimumab, breastfeeding should be discontinued if the mother is treated with LMB-100 + ipilimumab. These potential risks may also apply to other agents used in this study.
21. Human immunodeficiency virus (HIV) positive patients will be excluded due to a theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection.
22. Positive for Hepatitis B or C (defined as Hepatitis B surface antigen reactive) or known active Hepatitis C virus (defined as HCV ribonucleic acid (RNA) detected) infection. or active hepatitis B virus (HBV) or HCV infection.
23. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
24. Has an active infection requiring systemic therapy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data in Biomedical Translational Research Information System (BTRIS) will be shared throughout the course of the study and indefinitely with the permission of the investigator.
Access Criteria: Clinical individual participant data (IPD) will be shared through the Biomedical Translational Research Information System (BTRIS) database for open-ended analysis. All BTRIS subscribers, generally limited to the National Institutes of Health (NIH) Clinical Center, may request data.

REFERENCES:
- [Derived] Morhard R, Mauda-Havakuk M, Delgado JF, Kassin MT, Ghafoor A, Pastan I, Hassan R, Karanian JW, Pritchard WF, Wood BJ, Mikhail AS. Mapping drug distribution using CT imaging following direct tissue injection in ex vivo liver: informing clinical implementation. CVIR Oncol. 2025;1(1):27. doi: 10.1007/s44343-025-00027-x. Epub 2025 Dec 16. PMID 41425223
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000059-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level -1: 200 mcg LMB-100: Dose Level -1: 200 mcg LMB-100 administered per dose, dose administered on days 1 and 4 of 21-day cycle, cycle 1 in participants with pleural or peritoneal mesothelioma.
  Those with pleural or peritoneal mesothelioma receiving intra-tumoral administration of LMB-100 + Ipilimumab for up to 4 cycles.
  For infusion related reactions precaution, all participants will be premedicated 30-60 minutes (+ 30 minutes) prior to each LMB-100 administration with the following medications: Diphenhydramine 25-50 mg by mouth (PO) or intravenous (IV) (or alternative antihistamine at adequate dose), Famotidine 20 mg by mouth (PO) or intravenous (IV) (or alternative histamine H2- receptor antagonists (H2) blocker at adequate dose), and Acetaminophen 650 mg by mouth (PO) or intravenous (IV).
  Additional infusion precaution at infusions of LMB-100 after Cycle 1 Day 1 (as appropriate): Dexamethasone 20 mg by mouth (PO), 6-12 hours prior to LMB-100 administration OR 10mg, intravenous (IV), 30-60 minutes prior to LMB-100 administration OR equivalent dose of another corticosteroid as clinically indicated.
  Biopsy as feasible at screening, Cycle 1 Day 1 and 5, Cycle 2, 3, & 4 Day 1, and Cycle 4 Day 21 (±7 days).
- Dose Level 1: 400 mcg LMB-100: Dose Level 1: 400 mcg LMB-100 administered per dose, dose administered on days 1 and 4 of 21-day cycle, cycle 1 in participants with pleural or peritoneal mesothelioma.
  Those with pleural or peritoneal mesothelioma receiving intra-tumoral administration of LMB-100 + Ipilimumab for up to 4 cycles.
  For infusion related reactions precaution, all participants will be premedicated 30-60 minutes (+ 30 minutes) prior to each LMB-100 administration with the following medications: Diphenhydramine 25-50 mg by mouth (PO) or intravenous (IV) (or alternative antihistamine at adequate dose), Famotidine 20 mg by mouth (PO) or intravenous (IV) (or alternative histamine H2- receptor antagonists (H2) blocker at adequate dose), and Acetaminophen 650 mg by mouth (PO) or intravenous (IV).
  Additional infusion precaution at infusions of LMB-100 after Cycle 1 Day 1 (as appropriate): Dexamethasone 20 mg by mouth (PO), 6-12 hours prior to LMB-100 administration OR 10mg, intravenous (IV), 30-60 minutes prior to LMB-100 administration OR equivalent dose of another corticosteroid as clinically indicated.
  Biopsy as feasible at screening, Cycle 1 Day 1 and 5, Cycle 2, 3, & 4 Day 1, and Cycle 4 Day 21 (±7 days).
- Dose Level 2: 1200 mcg LMB-100: Dose Level 2: 1200 mcg LMB-100 administered per dose, dose administered on days 1 and 4 of 21-day cycle, cycle 1 in participants with pleural or peritoneal mesothelioma.
  Those with pleural or peritoneal mesothelioma receiving intra-tumoral administration of LMB-100 + Ipilimumab for up to 4 cycles.
  For infusion related reactions precaution, all participants will be premedicated 30-60 minutes (+ 30 minutes) prior to each LMB-100 administration with the following medications: Diphenhydramine 25-50 mg by mouth (PO) or intravenous (IV) (or alternative antihistamine at adequate dose), Famotidine 20 mg by mouth (PO) or intravenous (IV) (or alternative histamine H2- receptor antagonists (H2) blocker at adequate dose), and Acetaminophen 650 mg by mouth (PO) or intravenous (IV).
  Additional infusion precaution at infusions of LMB-100 after Cycle 1 Day 1 (as appropriate): Dexamethasone 20 mg by mouth (PO), 6-12 hours prior to LMB-100 administration OR 10mg, intravenous (IV), 30-60 minutes prior to LMB-100 administration OR equivalent dose of another corticosteroid as clinically indicated.
  Biopsy as feasible at screening, Cycle 1 Day 1 and 5, Cycle 2, 3, & 4 Day 1, and Cycle 4 Day 21 (±7 days).
Period: Overall Study
Arm/Group | Dose Level -1: 200 mcg LMB-100 | Dose Level 1: 400 mcg LMB-100 | Dose Level 2: 1200 mcg LMB-100
Started | 0 | 2 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 2 | 0
Not completed — None of the participants completed all 4 cycles. | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Intratumorally Administered LMB-100 in Participants With Mesothelioma
Description: RP2D is defined as the highest dose at which fewer than 2 of 6 participants experience a dose-limiting toxicity. A dose-limiting toxicity is defined as any Grade 4 hematological toxicity lasting greater than 5 days. Grade 3 febrile neutropenia, Grade 3 thrombocytopenia associated with bleeding episodes, any Grade 3 or greater, non-hematological toxicity with the following exceptions: tumor lysis syndrome, Grade 3 electrolyte changes associated with clinically significant consequences, Grade 3 nausea and diarrhea which has not received appropriate treatment, isolated Grade 3 fever occurring within 48 hours of LMB-100 infusion and resolving within 48 hours to ≤ Grade 2 and fully resolved within 1 week, alopecia, infusion-related reactions up to and including Grade 3, asymptomatic ≥ Grade 3 lymphopenia, leukopenia, hypoalbuminemia, electrolyte abnormalities resolving within 24 hours, and increase in alkaline phosphatase.
Time Frame: 21 days after first LMB-100 administration
Measure: Number; unit: mcg/kg
Groups:
- All Participants in Dose Level 1: 400 mcg LMB-100: All participants that received at least one dose of both LMB-100 and Ipilimumab.
  Dose Level 1: 400 mcg LMB-100 administered per dose, dose administered on days 1 and 4 of 21-day cycle, cycle 1 in participants with pleural or peritoneal mesothelioma.
  Those with pleural or peritoneal mesothelioma receiving intra-tumoral administration of LMB-100 + Ipilimumab for up to 4 cycles.
  For infusion related reactions precaution, all participants will be premedicated 30-60 minutes (+ 30 minutes) prior to each LMB-100 administration with the following medications: Diphenhydramine 25-50 mg by mouth (PO) or intravenous (IV) (or alternative antihistamine at adequate dose), Famotidine 20 mg by mouth (PO) or intravenous (IV) (or alternative histamine H2- receptor antagonists (H2) blocker at adequate dose), and Acetaminophen 650 mg by mouth (PO) or intravenous (IV).
  Additional infusion precaution at infusions of LMB-100 after Cycle 1 Day 1 (as appropriate): Dexamethasone 20 mg by mouth (PO), 6-12 hours prior to LMB-100 administration OR 10mg, intravenous (IV), 30-60 minutes prior to LMB-100 administration OR equivalent dose of another corticosteroid as clinically indicated.
Arm/Group | All Participants in Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
mcg/kg | NA — The RP2D was not determined because the study closed early due to lack of accrual.

2. Primary Outcome: Number of Participants Who Experienced Grades 1-5 Serious and/or Non-serious Toxicity Related (= Possibly + Probably + Definitely) to LMB-100
Description: Toxicity was assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. And Grade 5 is death related to adverse event.
Time Frame: Median follow-up: 3.4 months (1.9 months and 5.0 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
Participants
  Grade 1 Non-Serious Abdominal pain | 1
  Grade 1 Non-Serious Edema limbs | 1
  Grade 1 Non-Serious Fatigue | 1
  Grade 1 Non-Serious Hypoalbuminemia | 2
  Grade 1 Non-Serious Non-cardiac chest pain | 2
  Grade 1 Non-Serious Weight gain | 1
  Grade 2 Non-Serious Anemia | 1
  Grade 2 Non-Serious Capillary leak syndrome | 1
  Grade 2 Non-Serious Edema limbs | 1
  Grade 2 Non-Serious Hypoalbuminemia | 2
  Grade 2 Non-Serious Pneumonitis | 1
  Grade 2 Non-Serious Sinus tachycardia | 1
  Grade 3 Serious and/or Non-Serious Events | 0
  Grade 4 Serious Pericardial tamponade | 1
  Grade 5 Serious and/or Non-Serious Events | 0

3. Primary Outcome: Number of Participants Who Experienced Grades 1-5 Serious and/or Non-serious Toxicity Related (= Possibly + Probably + Definitely) to Ipilimumab
Description: as for outcome 2
Time Frame: Median follow-up: 3.4 months (1.9 months and 5.0 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
Participants
  Grade 1 Non-Serious Abdominal pain | 1
  Grade 1 Non-Serious Hypoalbuminemia | 1
  Grade 2 Non-Serious Hypoalbuminemia | 1
  Grade 2 Non-Serious Hypoxia | 1
  Grade 2 Non-Serious Pneumonitis | 1
  Grade 3 Serious and/or Non-Serious Events | 0
  Grade 4 Serious and/or Non-Serious Events | 0
  Grade 5 Serious and/or Non-Serious Events | 0

4. Secondary Outcome: Proportion of Participants Who Experienced an Objective Response Defined as Either a Partial or Complete Response
Description: Proportion of participants who experienced an objective response defined as either a partial or complete response assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Partial response is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Complete response is disappearance of all target lesions.
Time Frame: Median: 3.4 months (1.9 months and 5.0 months).
Measure: Number; unit: proportion of participants
Arm/Group | Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
proportion of participants
  Partial Response | 0
  Complete Response | 0

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the median time criteria are met for partial or complete response to the first date that recurrence or progression is documented. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Partial response is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Complete response is disappearance of all target lesions. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: Median follow-up: 3.4 months (1.9 months and 5.0 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
Months | NA [NA to NA] — Since participants had no response, we cannot provide duration of response.

6. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the median time from start of treatment to time of progression or death, whichever occurs first. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: Median: 1.4 months (95% CI: 0.6-2.3 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
Months | 1.4 [0.6 to 2.3]

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the median time from start of treatment to death from any cause.
Time Frame: Median 3.4 months (1.9 months and 5.0 months).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
Months | 3.4 [1.9 to 5.0]

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 7 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 400 mcg LMB-100
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 7 months.
Arm/Group | Dose Level 1: 400 mcg LMB-100
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 400 mcg LMB-100 (N=2)
Death NOS (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Pericardial tamponade (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 400 mcg LMB-100 (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (5)
Allergic reaction (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (4)
Fatigue (General disorders) | 2 (4)
Fever (General disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (16)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5)
Hypotension (Vascular disorders) | 2 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (11)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pericardial effusion (Cardiac disorders) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (6)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Thyroid stimulating hormone increased (Endocrine disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Weight gain (Investigations) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04840615/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT04840615/ICF_001.pdf